CLINICAL TRIAL: NCT03583021
Title: Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine
Brief Title: Sugammadex on Remifentanil Ce for Preventing Emergence Cough in Male
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-18-105
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Gallbladder Diseases
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sugammadex group (Experimental): Sugammadex group receives the intravenous sugammadex of 3 mg/kg.
  Interventions: Drug: Sugammadex Injectable Product
- neostigmine group (Placebo Comparator): Neostigmine group receives the intravenous neostigmine 50 ug/kg and glycopyrrolate 10 ug/kg.
  Interventions: Drug: Neostigmine Injectable Product

INTERVENTIONS:
Drug: Sugammadex Injectable Product — Sugammadex of 3 mg/kg is injected.
  Arms: sugammadex group
Drug: Neostigmine Injectable Product — Neostigmine of 50 ug/kg and Glycopyrrolate of 10 ug/kg are injected.
  Arms: neostigmine group

SUMMARY:
The primary purpose of this study is to investigate the optimal Ce of remifentanil for preventing emergence cough following extubation during general anesthesia in male patients who are reversed with sugammadex or neostigmine.

DETAILED DESCRIPTION:
Remifentanil is a potent ultrashort-acting opioid, with rapid onset and offset of drug effect. It allows rapid anesthetic emergence even after a prolonged infusion, and decreases the at-risk time during extubation. In addition, cough suppression of remifentanil enables smooth extubation with reduced complications. However, the infusion of remifentanil suppresses the emergence cough effectively in clinical practice, whereas it still delays the awakening from anesthesia, resulting in prolonged emergence time. Reduced Ce of remifentanil during emergence would decrease the adverse events that are associated with remifentanil infusion.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* BMI > 30 kg/m2, respiratory infection, uncontrolled hypertension

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
optimal Ce of remifentanil | from the ene of surgery until endotracheal extubation
  Using Dixon methods, evaluating of optimal Ce of remifentanil for preventing emergence cough following extubation during general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Ji Eun Kim, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoul, South Korea